CLINICAL TRIAL: NCT05999071
Title: Coriandrum Sativum Seeds Improve Memory, Alleviate Anxiety and Depression, and Enhance Sleep Quality in University Students: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hashemite University (Other)
Responsible Party: Principal Investigator, Abdelrahim Alqudah, Assisstant professor, The Hashemite University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 21/6/2022/2023
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Memory Disorders; Anxiety Depression; Sleep
Keywords: Coriandrum sativum; memory performance; anxiety; depression; sleep
MeSH Terms: conditions — Memory Disorders; Anxiety Disorders; Depression | interventions — coriander oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coriandrum sativum group (Experimental): 500 mg of C. sativum (capsules) were administered twice daily
  Interventions: Dietary Supplement: Coriandrum sativum seeds
- control group (Placebo Comparator): 500 mg of starch (capsules) were administered twice daily
  Interventions: Dietary Supplement: Coriandrum sativum seeds

INTERVENTIONS:
Dietary Supplement: Coriandrum sativum seeds — Each group consisted of 50 students. In the C. sativum group, dried powdered seeds of C. sativum were administered, while in the control group, starch was provided as a placebo. Both the C. sativum and placebo capsules were identical in shape, color, and outer packaging to maintain the blinding of the participants.
  Other Names: Coriandrum

SUMMARY:
C. sativum could potentially serve as a memory enhancer for university students. It is considered a preferable option to stimulant drugs due to its safety profile. Additionally, C. sativum may have positive effects on anxiety, depression, and sleep quality. However, it is important to note that the current body of research on the effects of oral C. sativum on the brain and nervous system is limited, and further studies are necessary to fully understand its potential benefits. Thus, this study aims to assess the impact of oral C. sativum on memory performance, anxiety, depression, and sleep quality in university students.

DETAILED DESCRIPTION:
Coriander, scientifically known as Coriandrum sativum L (C. sativum), is an ancient herb that belongs to the Apiaceae family. It has a rich history of more than 3,000 years of use in both culinary and medicinal practices. While originally native to Mediterranean regions, coriander is now cultivated in various countries worldwide. In traditional medicine, all parts of the coriander plant have been consumed and utilized to address gastrointestinal ailments like anorexia, dyspepsia, flatulence, diarrhea, pain, and vomiting. In Jordanian traditional medicine, C. sativum has been valued for its anticonvulsant, antidepressant, sedative, and anxiolytic properties. Studies have reported diverse health benefits associated with C. sativum seeds and leaves, including antioxidant, diuretic, cholesterol-lowering, anxiolytic, sedative-hypnotic, and anticonvulsant activities. Notably, the main component of C. sativum, linalool, along with γ-terpinene and α-pinene, exhibit various neuropharmacological effects, such as anti-anxiety, sedative, anticonvulsant, and anti-Alzheimer's disease properties. Additionally, C. sativum seeds are recognized as a valuable source of vitamins, lipids, and minerals like potassium, calcium, phosphorus, magnesium, sodium, and zinc.

Several studies have indicated the positive effects of C. sativum on memory, anxiety, and depression. In a specific study, the aqueous extract derived from the seeds of C. sativum demonstrated significant reductions in monoamine oxidase-B (MAO-B) activity over time, suggesting its primary role in exerting antidepressant-like effects. Another study reported that the administration of C. sativum leaves improved memory performance and hindered the aging process in rats in a dose-dependent manner. Furthermore, it was observed that C. sativum leaves reversed memory impairments induced by scopolamine and diazepam, while also significantly reducing brain cholinesterase activity and serum total cholesterol levels. Another study evaluated the effects of the ethanolic extract of C. sativum seeds on learning in second-generation mice. Although the plant extract did not enhance learning in the short term following training, it did show improvements in long-term learning. Additionally, in an animal model of anxiety, the effects of different doses (10 mg/kg, 25 mg/kg, 50 mg/kg, and 100 mg/kg administered intraperitoneally) of the aqueous extract of C. sativum seeds were evaluated in terms of motor activity and neuromuscular function. In the elevated plus-maze test, the 100 mg/kg dose of the seeds' aqueous extract exhibited anxiolytic effects by increasing the time spent in and the number of entries into the open arms.

Anxiety, depression, and sleep disorders are prevalent among university students, and these conditions can have a considerable impact on their memory function. Consequently, there has been a rise in the use of stimulant drugs among university students as a means to enhance memory performance and attention, despite the fact that such use is unapproved and non-therapeutic which might be associated with several side effects. As a result, there is a growing interest among neuroscience researchers to identify cognitive-enhancing drugs that can be safely used by healthy individuals without adverse effects.

Given the information provided, it is suggested that C. sativum could potentially serve as a memory enhancer for university students. It is considered a preferable option to stimulant drugs due to its safety profile. Additionally, C. sativum may have positive effects on anxiety, depression, and sleep quality. However, it is important to note that the current body of research on the effects of oral C. sativum on the brain and nervous system is limited, and further studies are necessary to fully understand its potential benefits. Thus, this study aims to assess the impact of oral C. sativum on memory performance, anxiety, depression, and sleep quality in university students.

ELIGIBILITY:
Inclusion Criteria:

* Male or female university Student.
* 19-23 of age

Exclusion Criteria:

* Medical diseases.
* Psychiatric disorders.
* Using any form of medication (including complementary and alternative medicines).
* Pregnant and lactating individuals.

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Memory performance | 30 days
  Prospective and Retrospective Memory Questionnaire was performed

SECONDARY OUTCOMES:
Anxiety and depression | 30 days
  Hospital Anxiety and Depression Scale was perfomed
Sleep quality | 30 days
  Pittsburgh Sleep Quality Inventory questionnaire was perfoemed

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmaceutical Sciences, Zarqa, Jordan

IPD SHARING:
Plan to Share IPD: No
All participants data will be hidden